CLINICAL TRIAL: NCT06698874
Title: Diagnostic Efficacy of Magnetically Controlled Capsule Endoscopy (MCE) for Identification of Bleeding Lesions in Patients with Antiplatelet Drugs-Related Acute Non-Hematochezia Gastrointestinal Bleeding：Prospective, Multicenter Study
Brief Title: MCE Identifying Bleeding Lesions in Patients with Antiplatelet Drugs-Related Acute Non-Hematochezia Gastrointestinal Bleeding
Acronym: MCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCTECT-BL
Record Dates: First submitted 2024-10-29; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Gastrointestinal Bleeding; Antiplatelet Therapy
Keywords: magnetically controlled capsule endoscopy; string; antiplatelet drugs; gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- group of participants (Experimental): Patients with antiplatelet drugs-related acute non-hematochezia gastrointestinal bleeding are enrolled. All enrolled participants will undergo the examination of detachable string magnetically controlled capsule endoscopy (ds-MCE) first, followed by EGD within 24 hours.
  Interventions: Other: ds-MCE and EGD examinations

INTERVENTIONS:
Other: ds-MCE and EGD examinations — Sequentially performing ds-MCE and EGD examinations on enrolled participants.

SUMMARY:
The goal of this clinical trial is to explore the diagnostic efficacy of detachable string magnetically controlled capsule endoscopy (ds-MCE) for identification of bleeding lesions in patients with antiplatelet drugs-related acute non-hematochezia gastrointestinal bleeding. The main questions it aims to answer are:

Compared to the conventional esophagogastroduodenoscopy, does ds-MCE accurately detect bleeding lesions in the upper gastrointestinal tract in patients with antiplatelet drugs-related acute non-hematochezia gastrointestinal bleeding? Recording bleeding lesions in the small bowel detected by ds-MCE in patients with antiplatelet drugs-related acute non-hematochezia gastrointestinal bleeding.

Participants will:

Undergo ds-MCE first and subsequently EGD within 24 hours. Receive follow-up in the following 30days.

DETAILED DESCRIPTION:
Antiplatelet therapy can effectively reduce the occurrence of thrombotic events, which is the primary treatment of cardiovascular and cerebrovascular diseases. However, long-term use of antiplatelet drugs can significantly increase the risk of gastrointestinal mucosal injury, and in severe cases can cause ulcers and bleeding. In patients with gastrointestinal bleeding related to antiplatelet drugs, it is crucial to identify the cause of bleeding, provide effective treatment and adjust antiplatelet treatment in time.

Hematemesis and melena are common clinical manifestations of upper gastrointestinal bleeding, as well as some patients with lower gastrointestinal bleeding.Previous studies have demonstrated that in patients taking long-term antiplatelet drugs, bleeding events occurred not only in the upper digestive tract but also in the lower digestive tract. For patients with hematemesis and melena, clinical guidelines recommend esophagogastroduodenoscopy (EGD) within 24 hours. When EGD fails to find bleeding lesions, clinical guidelines recommend further selection of colonoscopy, capsule endoscopy, enteroscopy, angiography and other methods to find bleeding lesions. However, EGD is invasive and there is potential for procedure-related complications. Besides, EGD can not further evaluate the small bowel, and small bowel mucosal lesions may be missed.

Ds-MCE has offered an noninvasive and safty modality for comprehensive examination of the upper digestive tract and small bowel.ds-MCE adds a detachable string to the conventional MCE, which can control the movement of the capsule through the string in the esophagus. In the process of stomach examination, the capsule position and direction is controlled under the external magnetic field. In the duodenum, ds-MCE can realize repeated observation of duodenum through the joint control of string and magnetic field. At the same time, the battery power of the capsule is longer than 8 hours, and the string can be separated from the capsule after the upper digestive tract examination. For patients with gastrointestinal bleeding undergoing antithrombotic therapy, ds-MCE is comfortable and non-invasive, and can complete upper gastrointestinal and small bowel examinations at one time, which is expected to improve the detection efficiency of bleeding lesions.

This study is a multicenter, prospective study. Patients with antiplatelet drugs-related acute non-hematochezia gastrointestinal bleeding were enrolled. Ds-MCE and EGD were performed successively. This study is aimed to evaluate the diagnostic efficacy of ds-MCE in the detection of bleeding lesions in patients with acute non-hematochezia gastrointestinal bleeding associated with antiplatelet drugs, using EGD as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. No gender limit, age ≥ 18 years；
2. Acute non-hematochezia gastrointestinal bleeding symptoms, including haematemesis or melena；
3. Taking antiplatelet drugs continuously for at least 14 days；
4. Hemodynamically stable；
5. Able to provide informed consent.

Exclusion Criteria:

1. Age < 18 years；
2. Hemodynamically unstable even after initial volume resuscitation and/or have ongoing fresh hematemesis at presentation；
3. With upper gastrointestinal bleeding caused by peptic ulcer or acute gastric mucosal lesion within 1 month before inclusion；
4. History of endoscopic therapy (such as ESD, EMR, etc.) within 1 month before inclusion；
5. Gastrointestinal tumor, decompensation of cirrhosis with esophageal or gastric varices；
6. Haematopathy and bleeding tendency；
7. Patients who have no surgical conditions or refuse to undergo any abdominal surgery (once the capsule is stuck, it cannot be removed surgically)；
8. Pacemaker or other implanted electromedical devices which could interfere with magnetic resonance；
9. Patients plan to undergo magnetic resonance imaging examination before excretion of the capsule；
10. Suspected or known intestinal stenosis or other known risk factors for capsule retention.
11. Pregnancy；
12. Dysphagia；
13. With and conditon contraindicated to ds-MCE or EGD；
14. With and conditon that is not suitable for participation in the study evaluated by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
the sensitivity and specificity of ds-MCE in detecting bleeding lesions in the upper gastrointestinal tract | from enrollment to the end of end of follow-up at 30 days
  the sensitivity and specificity of ds-MCE in identifying bleeding lesions in the upper gastrointestinal tract in patients with non-hematochezia gastrointestinal bleeding, using the detection by EGD as the reference standard.

SECONDARY OUTCOMES:
the diagnostic yield of ds-MCE in detecting bleeding lesions in the small bowel | from enrollment to the end of end of follow-up at 30 days
  the diagnostic yield of ds-MCE in identifying bleeding lesions in the small bowel in patients with antiplatelet drugs-related acute non-Hematochezia gastrointestinal bleeding
per-patient diagnostic yield of ds-MCE and EGD | from enrollment to the end of follow-up at 30 days
  diagnostic yield of ds-MCE and EGD in a per-patient analysis, using EGD as the reference standard in the upper gastrointestinal tract and MCE as the reference standard in the small bowel
gastrointestinal bleeding lesion detection rate of ds-MCE and EGD in a per-lesion analysis | from enrollment to the end of follow-up at 30 days
  gastrointestinal bleeding lesion detection rate of ds-MCE and EGD in a per-lesion analysis, using EGD as the reference standard in the upper gastrointestinal tract and MCE as the reference standard in the small bowel
endoscopy intervention rate | from enrollment to the end of follow-up at 30 days
  rate of participants who need further endoscopy intervention after ds-MCE
the examination time of ds-MCE and EGD | from enrollment to the end of follow-up at 30 days
  examination time of ds-MCE include esophageal transit time (ETT), gastric examination time (GET), gastric transit time (GTT), small bowel transit time (SBTT), and total running time (TRT).
comfort evaluation | from enrollment to the end of follow-up at 30 days
  patient comfort score of ds-MCE and EGD procedures
safety evaluation | from enrollment to the end of follow-up at 30 days
  all adverse events occurring during the study

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital
Locations (4):
- China (4):
  - Qinghai Special Hospital of Cardio-Cerebrovascular Disease, Qinghai
  - Changhai Hospital, Shanghai
  - Shanghai East Hospital, Tongji University School of Medicine, Shanghai
  - First Affiliated Hospital Xi'an Jiaotong University, Xi'an